CLINICAL TRIAL: NCT04268602
Title: The Effect of Intradermal Local Anesthetic Injection on Pain and Functionality in Failed Back Surgery Syndrome
Brief Title: The Effect of Intradermal Local Anesthetic Injection in FBSS (Failed Back Surgery Syndrome)
Acronym: FBSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Duygu Geler Külcü, Clinical Professor Dr, Head of Physical Medicine and Rehabilitation Department, Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HNEAH-KAEK2019/23-757
Record Dates: First submitted 2020-01-10; First posted 2020-02-13 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Failed Back Surgery Syndrome; Pain, Chronic
Keywords: FBSS; Failed Back Surgery Syndrome; Chronic Pain; local anesthetic; Intradermal Injection
MeSH Terms: conditions — Failed Back Surgery Syndrome; Chronic Pain | interventions — Anesthetics, Local; Exercise; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): intradermal 1% lidocain injection 4 cc+ exercise and transcutaneous electrical nerve stimulation
  Interventions: Other: local anesthetic injection
- Control Group (No Intervention): exercise and transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: local anesthetic injection — 1% lidocaine
  Other Names: exercise and transcutaneous electrical nerve stimulation
  Arms: Intervention Group

SUMMARY:
Failed Back Surgery Syndrome is described as chronic pain in the low back and/or legs after a spinal procedure. It is estimated that %10 - 40 of the patients who had spinal surgery will have Failed Back Surgery Syndrome. The aim of this study is to research whether intradermal injection of the local anesthetic on the operation scar area and the area in which pain referred to in patients with Failed Back Surgery Syndrome has effects on pain and functionality or not.

DETAILED DESCRIPTION:
The prevalence of low back pain is around 60% - 80% and its the 5th most common disease to seek medical help. 80% of patients who have an acute onset of low back pain whether treated or not relieved on symptoms, while unfortunately 10% of patients' low back pain will worsen end eventually progress to chronic low back pain. With the increase on the number of different techniques on spinal surgery, and an increase in the number of patients who had risk factors undergone spinal surgery caused an increase in the number of patients who had new complaints after surgery. The term Failed Back Surgery Syndrome describes new complaints or not enough ease on the complaints of a patient who had spinal surgery. Due to the variation of the criteria of assessment, it is noted that around 10% -40% of the patients who had spinal surgery will have Failed Back Surgery Syndrome.

Failed Back Surgery Syndrome is commonly described as pain in low back and/or legs with difficulty in daily activities. Pain might be radicular or localized to the low back, it might be mechanic or neuropathic in nature.

Some of the pathologies that cause Failed Back Surgery Syndrome are loss of height on the disc, arthrosis, spinal stenosis caused by the hypertrophy of the facet joints, recurrent disc herniation, arachnoiditis, central stenosis, epidural fibrosis, instability, pseudoarthrosis, and discitis.

Rehabilitation is one of the vital parts of the treatment of Failed Back Surgery Syndrome. After a detailed patient history and a complete physical examination, clinicians should create a rehabilitation program that aims improvements on pain, functionality, quality of life and activities of daily living and is tailored for the patient. It is shown that patients who undergo rehabilitation programs had improvements in physical functionality, posture, and difficulties with walking. Other conservative treatments include cognitive behavioral therapy and noninvasive injection techniques.

Literature shows that multifidus muscle is damaged and atrophied in the patients who had spinal surgery. Also, there is a correlation between functional impairment and atrophy. Usually, the muscles that control flexion and extension of the low back are weak in patients who have low back pain. Extensor muscles, especially the erector spinae muscle group are the posterior stabilisers of the vertebral colon. Loss of endurance and weakness of these muscles and low back pain have a correlation and strengthening these muscles will result in an improvement in low back pain.

Injections of local anesthetics on chronic pain syndromes are being used successfully for a long time. There are some examples of successful interventions on pelvic pain, myofascial pain syndrome and nonspecific chronic low back pain in the literature. While surgery is the first line of treatment in cases where the cause is the compromise of the neural structures or spinal instability, the pain will increase with recurrent surgery in other causes. Ligaments of the intervertebral disc complex which are innervated by the nociceptive neurons, facet joints, and paravertebral muscles are thought to be the reason for pain in Failed Back Surgery Syndrome. In a systemic review that took place in 2015; the superiority of injections done with saline, a mixture of steroids and local anesthetics and steroids alone for facet joints and epidural injection procedure was investigated. Investigators demonstrated that injection with local anesthetics alone was effective in treatment. Another systemic review in 2019 showed that injection of local anesthetics was effective and was superior to botulinum toxin A in the treatment of myofascial pain.

Intradermal injection of a drug is related to longer pharmacological effects compared to intramuscular and subcutaneous injections. Lidocaine antinociceptive, analgesic, anti-bacterial, anti-fungal, anti-viral, wound healing, releasing of endogen opioid effects were demonstrated. In the light of all the information above, the investigators wanted to research whether intradermal injection of the local anesthetic in patients with Failed Back Surgery Syndrome has effects on pain and functionality or not.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with failed back surgery syndrome
* 18-75 years of age
* visual analogue pain score> 4 to be

Exclusion Criteria:

* Mental problems
* Having a disease affecting the central nervous system or peripheral nervous system
* Fixation operation to the lumbar region
* Physical therapy in the lumbar region within the last 3 months
* Injection from the lumbar region in the last 3 months
* Lidocaine allergy
* Needle phobia.
* Wound, infection, allergy, burn-type lesions in the area to be injected
* Malignity history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Pain Scale scores | baseline, immediately after the intervention, 1 month
  Visual analog scale for measurement of pain. Minimum-maximum scores are 0-10. Higher scores mean worse outcome
Change in OSWESTRY Disability Index scores | baseline, immediately after the intervention, 1 month
  Low Back Pain Disability Questionnaire. Minimum-maximum scores are 0-100. Higher scores mean worse outcome

SECONDARY OUTCOMES:
Change in Hospital anxiety and depression scores | baseline, immediately after the intervention, 1 month
  anxiety and depression evaluation. Minimum-maximum scores are 0-21. Higher scores mean worse outcome
change in modified schober test measurement | baseline, immediately after the intervention, 1 month
  measurement to asses the mobility of lumbar vertebrae (cm)
change in Lateral hand to ground test measurement | baseline, immediately after the intervention, 1 month
  measurement to asses the mobility of lumbar vertebrae (cm)

IPD SHARING:
Plan to Share IPD: No